CLINICAL TRIAL: NCT03049826
Title: Nutritional Status in Children Treated With Advanced Nutrition Therapy
Acronym: NUTRIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Christine Henriksen, Assossiate Professor, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AEV2017/1
Record Dates: First submitted 2017-02-01; First posted 2017-02-10 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Body Composition; Children
Keywords: nutrient
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stem cell transplantation (SCT) (Experimental): Children undergoing stem cell transplantation (SCT)
  Interventions: Other: Nutritional status
- Home parenteral nutrition (HPN) (No Intervention): Children receiving home parenteral nutrition
- Healthy reference group (No Intervention): Healthy children

INTERVENTIONS:
Other: Nutritional status — Body composition and nutrient status
  Arms: Stem cell transplantation (SCT)

SUMMARY:
Background: There are few studies about nutrition to children and adolescents with cancer, and in particular during stem cell transplantation (SCT). Studies from other countries suggest that malnutrition is common on admission; the situation decline during treatment and may persist for a long time.

Aim: This project aims to improve the nutritional therapy to children being treated for cancer and children undergoing stem cell transplantation

DETAILED DESCRIPTION:
Design, methodology and selection: The study consist of two parts: A retrospective study (registry study) of malnutrition among all children with cancer, admitted during a two year period, and a clinical trial to evaluate the effect of a standardized nutrition protocol for children undergoing SCT. Nutritional status is assessed before, during and one year after treatment with SCT.

The subjects are 140 children and adolescents (2-17 years) being treated for cancer and a subgroup of 25 patients treated with SCT at Oslo University. The results will be compared with a reference group of 25 patients treated with home parenteral nutrition as well as 50 healthy reference persons in the same age group.

The methods used for measurement of nutritional status are: Body composition, bone density, blood tests, diet record, activity detection and measurement of quality of life. The measurements are done on three occasions for patients with cancer and stem cell transplantation, and on one occasion with a reference. Information on demographics and medical care will be taken from journal. Growth data will be collected from health centres when needed. Parents' experiences of children's feeding problems will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be recruited from Oslo University Hospital. Inclusion criteria are age 2 -17 years of age. The SCT and HPN group will include children who have not previously undergone transplantation, who do not have a pacemaker or other implants that prevent the measurement of muscle mass. Participants in the reference groups will be of the same age group, without congenital syndromes or previous cancers.

Exclusion Criteria:

* Exclusion criteria are patients who reject bone marrow

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Body composition meassured with Lunar Dxa | After one year

SECONDARY OUTCOMES:
Blood vitamins and minerals | After one year
Dietary intake | After one year
Physical activity | After one year
Health related Quality of life | After one year

CONTACTS AND LOCATIONS:
Overall Officials: Christine Henriksen, PhD, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - University of Oslo, Oslo
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No